CLINICAL TRIAL: NCT01372306
Title: Comparative, Randomized, Single-Dose, 2-way Crossover Bioavailability Study of Dr.Reddy's Laboratories, Ltd. and Janssen Pharmaceutical Products, l.P. (Reminyl®)4 mg Galantamine HBr Tablets in Healthy Adult Male Volunteers Under Fed Conditions
Brief Title: Galantamine Bioequivalence Study of Dr. Reddy's Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Assistant Manager - Research & Development, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AA21897
Record Dates: First submitted 2011-01-27; First posted 2011-06-13 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2004-10

CONDITIONS: Fed
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency | interventions — Galantamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Galantamine (Experimental): Galantamine Hydrobromide Tablets of Dr. Reddy's
  Interventions: Drug: Reminyl
- Reminyl (Active Comparator): Reminyl 4 mg tablets of Janssen Pharmaceutical Products
  Interventions: Drug: Reminyl

INTERVENTIONS:
Drug: Reminyl — Galantamine Hydrobromide Tablets of Dr. Reddy's Laboratories Limited
  Other Names: Reminyl 4 mg

SUMMARY:
Galantamine Hydrobromide Tablets, Bioequivalence study of Dr. Reddy's under Fed condition.

DETAILED DESCRIPTION:
Comparative, Randomized, Single-Dose, 2-way Crossover Bioavailability Study of Dr.Reddy's Laboratories, ltd. and Janssen Pharmaceutical Products, l.P. (Reminyl®)4 mg Galantamine HBr Tablets in Healthy Adult Male Volunteers under Fed Conditions

ELIGIBILITY:
Inclusion Criteria:

Subject candidates must fulfill all of the following inclusion criteria to be eligible for participation in the studyI unless otherwise specified:

* Healthy adult male volunteers, 18-55 years of age;
* Weighing at least 60 kg and within 15% of their ideal weights (Table of "Desirable Weights of Adults", Metropolitan Ufe Insurance Company, 1983);
* Medically healthy subjects with clinically normal laboratory profiles, vital signs and ECGs;
* Give voluntary written informed consent to participate in the study.

Exclusion Criteria:

Subject candidates must not be enrolled in the stUdy if they meet any of the following criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease.
* In addition, history or presence of:
* alcoholism or drug abuse within the past year;
* hypersensitivity or idiosyncratic reaction to galantamine or other anticholinesterase inhibitors;
* asthma and seizures.
* Subjects who tested positive at screening for HIV, HbsAg or HCV.
* Subjects whose PR interval is >200 msec at screening and prior to dosing.
* Subjects whose QTc interval is >450 msec at screening and prior to dosing.
* Subjects who have used any drugs or substances known to be strong inhibitors of CYP enzymes (formerly known as cytochrome P450 enzymes) within 28 days prior to the first dose.
* Subjects who have used any drugs or substances known to be strong inducers of CYP enzymes (formerly known as cytochrome P450 enzymes) within 28 days prior to the first dose.
* Subjects who have been on a special diet (for whatever reason) during the 28 days prior to the first dose and throughout the study.
* Subjects who, through completion of the stUdy, would have donated in excess of:

  500 mL of blood in 14 days; 1500 mL of blood in 180 days; 2500 mL of blood in 1 year.
* Subjects who have participated in another clinical trial within 28 days prior to the first dose.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2004-10; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence on Cmax and AUC parameters | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Gaerano Morelli, Principal Investigator — Early Clinical Research